CLINICAL TRIAL: NCT07406984
Title: A Phase I Clinical Study to Evaluate the Safety and Efficacy of IM96 CAR-T Cell Injection in Advanced Adenocarcinoma of Gastric/Esophagogastric Junction
Brief Title: Clinical Study of IM96 CAR-T Cell Therapy in Patients With Advanced Adenocarcinoma of Gastric/Esophagogastric Junction
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMSZ9603
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Adenocarcinoma of Gastric/Esophagogastric Junction
Keywords: Advanced adenocarcinoma of gastric/esophagogastric junction IM96 CAR-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM96 CAR-T Cells (Experimental): After preconditioning with chemotherapy, IM96 CAR-T Cells will be evaluated
  Interventions: Biological: IM96 CAR-T Cells

INTERVENTIONS:
Biological: IM96 CAR-T Cells — IM96 CAR-T Cells, 6×10^8 CAR-T cells, 12×10^8 CAR-T cells, 20×10^8 CAR-T cells, treatment follows a lymphodepletion.Drug: Fludarabine Recommendation: 30 mg/m^2 (D-5~D- 3), determined by tumor burden at baseline.Drug: Fludarabine Recommendation: 30 mg/m^2 (D-5~D-3), determined by tumor burden at baseline.Drug:Cyclophosphamide Recommendation: 300mg/ m^2 (D-5~D-3), determined by tumor burden at baseline.

SUMMARY:
This study, a single-center, open, single-dose clinical study, was designed to evaluate the safety and efficacy of IM96 CAR-T cells in treating patients with advanced adenocarcinoma of gastric/esophagogastric junction

DETAILED DESCRIPTION:
This study is planned to enroll 18-24 patients with advanced adenocarcinoma of gastric/esophagogastric junction,using a modified "3+3" design for dose escalation, with 3 dose groups of 6×10^8 CAR-T cells ,12×10^8 CAR-T cells and 20×10^8 CAR-T cells. 3-6 subjects are planned to be enrolled in each dose group to assess their safety, and if the incidence of horizontal dose-limiting toxicity (DLT) is ≤1/6 within 28 days after transfusion in one dose group, the next dose group can be started. If the incidence of horizontal dose-limiting toxicity (DLT) in a dose group is ≤1/6 within 28 days after transfusion, transfusion of cells from the next dose group can be initiated.

This study will be divided into a screening period, a cell collection period, a chemotherapy pretreatment period, a return infusion and a follow-up period, and within 28 days of return infusion the investigator will assess whether a DLT (Dose limited toxicity) event has occurred to confirm the safety of this dose group.

ELIGIBILITY:
Inclusion Criteria:

1. The age is 18 to 75 years (including boundary values) and the gender is not limited;
2. Patients with advanced locally inoperable or metastatic adenocarcinoma of the stomach/gastric esophageal junction diagnosed by pathohistology;
3. Patients with metastatic stomach/gastric esophageal junction who have failed or are intolerant to standard therapy;

   Notes:
   1. The standardized systemic treatment received by the patient must be in accordance with the Chinese Society of Clinical Oncology (CSCO) Guidelines for the Treatment of Gastric Cancer, 2025 Edition;
   2. The standard prior treatment regimen should incorporate therapeutic strategies guided by relevant molecular biomarkers. Specifically, patients with HER2-positive tumors must have received HER2-targeted therapy;
   3. Claims of treatment intolerance: Patients who are unable to continue current effective systemic standardized treatment due to toxic side effects such as grade ≥3 vomiting, diarrhea, abdominal pain, bone marrow suppression, etc., and who do not accept refusal for financial and personal reasons;
4. Presence of at least one measurable lesion that meets RECIST 1.1 criteria;
5. Patients must provide a tumor sample within 2 years that meets the requirements (paraffin block or number of unstained sections that meet the testing requirements set by the Institute) that is positive for GUCY2C expression by immunohistochemistry;
6. Eastern cooperative oncology group (ECOG) score of 0-1;
7. Women of childbearing potential who have a negative blood pregnancy test prior to the start of the trial and who agree to use effective contraception during the trial and up to the last follow-up visit;male patients whose partners are of childbearing potential agree to use effective contraception during the trial and up to the last follow-up visit;
8. Laboratory tests should meet at least the indicators specified below:

   Hemoglobin (Hb) ≥ 80 g/L; Neutrophil count (Absolute neutrophil count, ANC) ≥ 1.5 x 10^9/L; Platelet count (PLT) ≥ 75 x 10^9/L; Absolute lymphocyte value ≥ 0.6 x 10^9/L; Lymphocytes make up ≥10% of white blood cells; Creatinine clearance ≥60 ml/min; Alanine transaminase (ALT) and Aspartate aminotransferase (AST) ≤ 2.5 x ULN and total bilirubin (TBL) ≤ 1.5 x ULN (for elevations of ALT and AST that can be explained by hepatic aggression, the high limits for AST and ALT can be adjusted upward to 5-fold, and the high limit for TBL may be adjusted upward to 3-fold; Serum albumin ≥ 3.0 g/dL; Prolongation of prothrombinogen time ≤ 4s;
9. Left ventricular ejection fraction ≥ 50% with a normal ECG or an abnormal ECG that, in the judgment of the investigator, does not require treatment;
10. Oxygen saturation >92% in non-oxygenated state;
11. Vascular access is adequate for cell collection, and lines are available for patients with existing central venous catheters;
12. Those who voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. Presence of brain metastases;
2. Patients who have previously received or are awaiting an organ transplant;
3. Toxicity due to prior therapy not stabilized or recovered to ≤ grade 1 (except in cases judged by the investigator to be not clinically significant);
4. Plasmapheresis (e.g., pleural effusion, abdominal effusion, pericardial effusion) with symptoms of compression that cannot be controlled with treatment;
5. Autoimmune disease requiring systemic immunosuppressive therapy (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus) within 2 years prior to the start of screening;
6. Lung diseases that the inversgaters determined were not suitable for inclusion in the study;
7. Use of any of the following medications or treatments during the designated time period prior to cell collection:

   1. Therapeutic doses of corticosteroids have been used within 7 days prior to cell collection. However, topical and inhaled steroids are permitted;
   2. Received chemotherapeutic agents within 1 week prior to cell collection. Enrollment was allowed if the oral chemotherapeutic drug had passed at least 3 half-lives prior to cell collection;
   3. Those who used drugs to stimulate bone marrow hematopoietic cell production within 5 days prior to cell collection;
   4. Use of study drug within 4 weeks prior to cell collection.However, enrollment was allowed if the trial treatment was ineffective or the disease progressed during the trial and at least 5 half-lives had elapsed prior to cell collection;
   5. Received interventional therapy, radiotherapy, ablation, and other localized treatments for the study disease within 4 weeks prior to cell collection;
   6. Patients who have had major surgery or significant trauma within 4 weeks prior to cell collection or who are expected to require major surgery during the study period;
   7. Received targeted drug treatment such as apatinib or fuyiquatine within one week prior to cell collection;
   8. Received immunotherapy drugs such as anti-PD-1/PD-L1 within four weeks prior to cell collection;
8. Prior treatment with anti-GUCY2C target (unless GUCY2C target test remains positive);
9. Those who have received other cell therapy or genetically modified cell therapy in the past, such as TCR-T therapy, CAR-T therapy, etc;
10. Prior or clinically significant CNS disorders at screening, such as epilepsy, epileptic seizures, cerebrovascular disease (ischemia/hemorrhage/cerebral infarction), cerebral edema, reversible posterior leukoencephalopathy, paralysis, aphasia, stroke, severe brain injury,dementia, Parkinson's disease, cerebellar disorders, organic brain syndromes, or psychiatric disorders;
11. Chronic or active infection requiring systemic therapy and history of symptomatic viral infection that has not been completely cured. For example, Hepatitis B: patients who are positive for Hepatitis B surface antigen (HBsAg) and/or Hepatitis B core antibody (HBcAb) and whose peripheral blood HBV-DNA test is above the lower limit of detection;patients who are positive for Hepatitis C Virus Antibody (HCVAb) and whose peripheral blood HCV-RNA test is above the lower limit of detection; and patients infected with Human Immunodeficiency Virus (HIV), Syphilis;
12. Active EBV and cytomegalovirus, defined as patients with IgM antibodypositive or IgM antibody-negative but higher-than-normal EBV-DNA in EBV serum; and cytomegalovirus (CMV) seropositive or IgM antibodynegative but higher-than-normal CMV-DNA in serum;
13. Vaccination with live vaccine within 6 weeks prior to the start of screening;
14. Abnormalities of cardiac function include: long QTc syndrome or QTc interval >480 ms; complete left bundle branch block, degree II/III AV block; severe, uncontrolled arrhythmias requiring pharmacologic therapy; history of chronic congestive heart failure with NYHA class ≥3 (refer to Attachment 3) with a cardiac ejection fraction of less than 50% in the 6 months prior to screening; CTC AE ≥3 grade heart valve disease;myocardial infarction, cardiac angioplasty or stenting,unstable angina, history of severe pericardial disease, or other clinically significant cardiac disease within 6 months prior to screening;
15. Patients requiring anticoagulation therapy;
16. Requires long-term use of medications that can affect clotting (e.g.,aspirin, warfarin, etc.);
17. History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months prior to initiation of screening;
18. Other untreated malignant tumors within the previous 5 years or concurrently, except cervical cancer in situ, basal cell carcinoma of the skin, and ductal carcinoma in situ of the breast;
19. Infections (fungal, bacterial, viral, or other) that require intravenous antimicrobial control or are uncontrollable, for simple urinary tract infections, and for bacterial pharyngitis, may be enrolled if the investigator evaluates that they can be controlled by curative treatment;
20. Patients with digestive tract obstruction;
21. The primary lesion exhibits a large ulcer, conferring a high risk of hemorrhage or perforation; alternatively, imaging studies (CT or MRI), with or without adjunctive gastroscopy, demonstrate transmural tumor invasion-i.e., infiltration across the full thickness of the gastric wall-thereby elevating the patient's risk of hemorrhage or perforation;
22. Patients present with unstable or active peptic ulcers, active gastrointestinal bleeding, or a history of major gastrointestinal bleeding within the preceding three months;
23. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study;
24. The presence of any factors affecting compliance with the protocol or the patient's unwillingness or inability to comply with the procedures required in the study protocol, as determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-03-05 (Estimated); Primary Completion 2027-05-05 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs) | Up to 28 days after CAR-T cell infusion
  Incidence of adverse events associated with IM96 CAR-T cell infusion within 28 days of IM96 CAR-T cell infusion,type, frequency, and severity of abnormal clinically significant vital signs, electrocardiograms, and laboratory tests examined, including dose-limiting toxicity

SECONDARY OUTCOMES:
Objective remission rate (ORR) | At 28 days, 3 months, 6 months and 12 months after CAR-T cell infusion
  Objective remission rate (ORR) after infusion
Progression-free survival (PFS) | At 28 days, 3 months, 6 months and 12 months after CAR-T cell infusion
  Progression-free survival (PFS) after infusion
Disease control rate (DCR) | At 28 days, 3 months, 6 months and 12 months after CAR-T cell infusion
  Disease control rate (DCR) after infusion
Duration of response (DOR) | At 28 days, 3 months, 6 months and 12 months after CAR-T cell infusion
  Duration of response (DOR) after infusion
Overall survival (OS) | At 28 days, 3 months, 6 months and 12 months after CAR-T cell infusion
  Overall survival (OS) after infusion
AUC (Area Under Curve) 0-D90 | Up to 90 days after CAR-T cell infusion
  AUC 0-D90 of IM96 CAR-T cells in vivo (peripheral blood) after infusion
Cmax (Peak Concentration) | Up to 28 days after CAR-T cell infusion
  Peak Concentrationof IM96 CAR-T cells in vivo (peripheral blood) after infusion
Tmax (Peak Time) | Up to 28 days after CAR-T cell infusion
  Peak Time of IM96 CAR-T cells in vivo (peripheral blood) after infusion
Tumor markers CA19-9 | At 28 days, 3 months, 6 months and 12 months after CAR-T cell infusion
  The changes of tumor markers CA19-9 before and after IM96 CAR-T cell infusion
Tumor markers CEA | At 28 days, 3 months, 6 months and 12 months after CAR-T cell infusion
  The changes of tumor markers CEA before and after IM96 CAR-T cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No